CLINICAL TRIAL: NCT07001540
Title: Evaluation of the Efficacy and Safety of Polatuzumab Vedotin Combined With Rituximab, Gemcitabine, and Oxaliplatin (Pola-R-GemOx) as Salvage Therapy for Relapsed/Refractory Diffuse Large B-Cell Lymphoma (DLBCL) Patients Ineligible for Autologous Transplantation: A Prospective, Multicenter, Single-Arm Clinical Study
Brief Title: Evaluation of the Efficacy and Safety of Polatuzumab Vedotin Combined With Rituximab, Gemcitabine, and Oxaliplatin (Pola-R-GemOx) as Salvage Therapy for Relapsed/Refractory Diffuse Large B-Cell Lymphoma (DLBCL) Patients Ineligible for Autologous Transplantation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: Fujian Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Rong Tao, Associate Chief Physician, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pola-R-Gemox
Record Dates: First submitted 2025-05-25; First posted 2025-06-03 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Diffuse Large B-Cell Lymphoma
Keywords: Polatuzumab vedotin combined with rituximab, gemcitabine and oxaliplatin (Pola-R-GemOx); Recurrent/refractory diffuse large B-cell lymphoma that is not suitable for autologous migration; Prospective, multicenter, single-armed
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Recurrence | interventions — Rituximab; Gemcitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment group (Experimental): Second-line salvage therapy for relapsed/refractory DLBCL patients ineligible for autologous transplantation.
  Interventions: Drug: Polatuzumab Vedotin combined with Rituximab, Gemcitabine, and Oxaliplatin (Pola-R- GemOx)

INTERVENTIONS:
Drug: Polatuzumab Vedotin combined with Rituximab, Gemcitabine, and Oxaliplatin (Pola-R- GemOx) — Polatuzumab Vedotin combined with Rituximab, Gemcitabine, and Oxaliplatin (Pola-R-GemOx)

SUMMARY:
This is a prospective, multicenter, single-arm clinical study designed to evaluate the efficacy and safety of Polatuzumab Vedotin combined with Rituximab, Gemcitabine, and Oxaliplatin (Pola-R-GemOx) as salvage therapy for relapsed/refractory Diffuse Large B-Cell Lymphoma (DLBCL) patients ineligible for autologous transplantation.

DETAILED DESCRIPTION:
This prospective, multicenter, single-arm Phase II clinical trial is designed to evaluate the efficacy and safety of Pola-R-GemOx in patients with relapsed/refractory diffuse large B-cell lymphoma (DLBCL) who are unsuitable for autologous transplantation. The study aims to enroll 130 patients, all of whom will initially receive three cycles of Pola-R-GemOx. Subsequent treatment decisions will be based on therapeutic efficacy and transplant assessment. ① Patients achieving complete response (CR) or partial response (PR) after three cycles will proceed with an additional three cycles. Those achieving CR following six cycles will conclude treatment, while all other patients will transition to subsequent-line therapy. ② Patients who do not achieve CR or PR after three cycles will discontinue the regimen and proceed directly to subsequent-line therapy. The primary endpoint of the trial is the investigator-assessed objective response rate (ORR). Secondary endpoints include other efficacy measures, such as complete response rate (CR), event-free survival (EFS), 24-month progression-free survival (PFS) rate, overall survival (OS), and safety outcomes. Additionally, exploratory analyses will be conducted to identify potential predictors of clinical efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

-

Participants must meet all of the following criteria to participate in the study:

1. Age ≥18 years old;
2. ineligible for autologous transplantation;
3. Sign the Informed Consent Form (ICF);
4. CD79b-positive DLBCL confirmed by pathology (including transformed DLBCL, PMBL, HGBCL);
5. Patients must have received adequate first-line treatment and only first-line treatment, with

   * Anti-CD20 monoclonal antibodies (unless the investigator determines that the tumor is CD20-negative)
   * Chemotherapy regimens containing anthracyclines
6. Recurrent or refractory diseases after first-line immunochemotherapy:

   * Refractory disease is defined as not having a complete response to first-line therapy (except for patients who are intolerant to first-line therapy)
   * Recurrent disease is defined as disease recurrence after complete response to first-line treatment
7. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2, with an expected survival of more than 12 weeks.
8. Have at least one measurable two-dimensional lesion identified by clinical examination, CT scan or MRI: ① lymph node >1.5cm; ② Other non-lymph node lesions ≥1.0cm;
9. The main tissues and organs function well:

Hematological function: absolute granulocyte count ≥ 1,000/mm3, platelet count ≥ 75,000/mm3; Liver function: ALT/AST < 3 times upper limit of normal (ULN) and total bilirubin ≤1.5× upper limit of normal (ULN) (< 5 times ULN in patients with Gilbert syndrome, cholestasis due to hilar compression adenopathy, biliary obstruction due to liver involvement or lymphoma); Renal function: creatinine clearance > 30 mL/min, creatinine ≤1.5× upper limit of normal (ULN) Lung function: indoor oxygen saturation ≥95%; Cardiac function: no obvious cardiac insufficiency or cardiovascular disease; 10. Fertile patients must be willing to use highly effective contraception during the study period and for 120 days after the last dose of treatment.

Exclusion Criteria:

-

Subjects who meet any of the following criteria are not eligible to participate in this study:

1. Subjects with any factor that may affect their ability to comply with the protocol, as determined by the investigator, including uncontrollable medical, psychological, family, social, or geographical conditions, or those unwilling or unable to follow the procedures required by the study protocol.
2. Known human immunodeficiency virus (HIV) infection or immunoassay positive；
3. Viral infections that cannot be controlled by antiviral drugs, such as active herpes virus infection, acute or chronic active hepatitis B, acute or chronic active hepatitis C, etc. (Note: chronic HBV carriers or inactive HBsAg positive subjects with HBV-DNA lower than the lower limit of detection can be enrolled, requiring clinical evaluation and preventive antiviral therapy if appropriate; HCV antibody negative can be enrolled, HCV antibody positive patients need to test HCV-RNA, if negative can be enrolled)
4. Patients with uncontrolled lymphomas with CNS infiltration (CNS disease diagnosed at initial diagnosis is allowed, provided complete remission of CNS disease is achieved and maintained and no CNS disease is present at recurrence);
5. Patients who have previously received oxaliplatin or gemcitabine treatment;
6. Pregnant or lactating patients;
7. Other concurrent serious illness or medical condition that would prevent participation in the study;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-05-08 (Actual); Primary Completion 2027-11-15 (Estimated); Study Completion 2027-11-15 (Estimated)

PRIMARY OUTCOMES:
Invetigator-assessed Objective Response Rate (ORR) | Assessed up to 3 years
  Defined as the proportion of all analyzable subjects achieving complete response (CR) and partial response (PR) after study initiation.

SECONDARY OUTCOMES:
The CR rate assessed by the investigator | Assessed up to 3 years
  Defined as the proportion of all analyzable subjects achieving complete response (CR) after study initiation.
Event-free survival (EFS) | Assessed up to 3 years
  Defined as the time from the start of treatment to disease progression/recurrence, death from any cause, or the start of next line lymphoma therapy (NALT); Patients who had not experienced an event at the time of analysis were excluded from the most recent disease assessment date.
24-month progression-free survival (PFS) rate | Assessed up to 24 months
  PFS is defined as the time between the start of treatment and first recording to disease progression or death; Patients who had not experienced an event at the time of analysis were excluded from the most recent disease assessment date.
Overall survival time (OS) | Assessed up to 15 years
  Defined as the time from the start of treatment until death from any cause; Patients who had not experienced an event at the time of analysis were deleted on the date the patient was last known to be alive.
Security | Assessed up to 3 years
  The incidence of adverse events (AES), defined as all adverse events that occurred after a patient received the investigatory treatment regimen; The incidence of treatment-related AES was defined as the incidence of AEs associated with salvage therapy, transplantation, and consolidation therapy considered by the investigator after a patient received the investigational treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Wenhao Zhang, M.D, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No